CLINICAL TRIAL: NCT01063413
Title: Impact Analysis of Metro Parks' After-School Programming on Physical Activity, Weight and Fitness Outcomes
Brief Title: Physical Activity, Weight and Fitness Outcomes in Children in After-Care
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 090986
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-01

CONDITIONS: Obesity; Exercise
Keywords: Behavioral Research; Community-Based Participatory Research
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Coleman Afterschool Program: Children enrolled in a community center-based after-school program.
- YMCA Fun Company: Children enrolled in a school-based after-school program.

SUMMARY:
The purpose of this study is to compare the effect of two after-school programs on children's physical activity, fitness, body composition, and academic performance.

DETAILED DESCRIPTION:
Tennessee ranks 4th for the highest prevalence of adult obesity in the nation (30.2%), and ranks 5th for the highest rate of youth obesity (36.5%). The Division of General Pediatrics at Vanderbilt has a specific research focus to develop community engagement projects that measurably reduce childhood obesity. Metro Parks and Recreation has been showcased by the National Recreation and Parks Association (NRPA) as a national model for its leadership role in community health and wellness. The two have created a unique academic-community partnership, guided by principals of community-based participatory research (CBPR), that is working to test and disseminate effective Metro Parks-based programs to reduce pediatric obesity. The proposed study will examine the impact of the Coleman Community Center after-school program on routine physical activity, weight and fitness outcomes in children who belong to the low-income and racial and ethnic minority populations at highest risk for childhood obesity. This study was requested by Metro Parks and has significant policy implications: If the program is deemed effective in improving daily physical activity, weight and/or fitness outcomes in students, the proposed study will serve as the rationale to expand the program to Metro Parks' 22 community centers, all of which are located in under-resourced neighborhoods.

ELIGIBILITY:
Inclusion Criteria:

* 5 - 15 years
* enrolled in public school district
* parental permission to access school records

Exclusion Criteria:

* under 5 or over 15
* no parental permission to access school records

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: public school students
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Physical activity measured by actigraphy | 3 weeks over 3 months

SECONDARY OUTCOMES:
Body composition measured by bioelectrical impedance | 3 times over 3 months
Cardiovascular fitness measured by 1/2 mile run/walk | 3 times over 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sabina B. Gesell, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Metro Parks & Recreation - Coleman Park Regional Center, Nashville, Tennessee
  - YMCA Fun Company - Glencliff Elementary School, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
These data have been shared with researchers who have contacted the PI, Dr. Sabina Gesell at sgesell@wakehealth.edu.

REFERENCES:
- [Result] Gesell SB, Tesdahl E, Ruchman E. The distribution of physical activity in an after-school friendship network. Pediatrics. 2012 Jun;129(6):1064-71. doi: 10.1542/peds.2011-2567. Epub 2012 May 28. PMID 22641755
- [Result] Gesell SB, Sommer EC, Lambert EW, Vides de Andrade AR, Whitaker L, Davis L, Beech BM, Mitchell SJ, Arinze N, Neloms S, Ryan CK, Barkin SL. Comparative effectiveness of after-school programs to increase physical activity. J Obes. 2013;2013:576821. doi: 10.1155/2013/576821. Epub 2013 Aug 4. PMID 23984052
- [Result] Zhang J, Shoham DA, Tesdahl E, Gesell SB. Network interventions on physical activity in an afterschool program: an agent-based social network study. Am J Public Health. 2015 Apr;105 Suppl 2(Suppl 2):S236-43. doi: 10.2105/AJPH.2014.302277. Epub 2015 Feb 17. PMID 25689202
- [Result] Henry T, Gesell SB, Ip EH. Analyzing heterogeneity in the effects of physical activity in children on social network structure and peer selection dynamics. Netw Sci (Camb Univ Press). 2016 Sep;4(3):336-363. doi: 10.1017/nws.2016.2. Epub 2016 May 12. PMID 27867518